CLINICAL TRIAL: NCT05664269
Title: The Evaluation of Canola Protein and Whey Protein to Support Muscle Conditioning in Vivo in Young Females
Brief Title: Anabolic Properties of Canola
Acronym: ALPACA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Maastricht University Medical Center (Other)
Collaborators: DSM Food Specialties (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: NL81203.068.22 / METC 22-031
Record Dates: First submitted 2022-11-22; First posted 2022-12-23 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2022-12

CONDITIONS: Muscle Protein Synthesis
Keywords: Dietary protein; resistance exercise; Plant protein; muscle metabolism
MeSH Terms: interventions — Dietary Supplements; Resistance Training

STUDY DESIGN:
Intervention Model Description: randomized, controlled, parallel-group, double-blind intervention trial.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Randomization of interventional drinks will be performed by an independent researcher who will also prepare the drinks on the morning of the test day. Drinks will be prepared in a non-transparent shaker and matched for taste.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Canola protein (Experimental): 20g of canola protein
  Interventions: Dietary Supplement: drink ingestion; Behavioral: resistance-type exercise
- Whey protein (Active Comparator): 20g of whey protein
  Interventions: Dietary Supplement: drink ingestion; Behavioral: resistance-type exercise
- Placebo (Sham Comparator): Water, matched for taste and volume
  Interventions: Dietary Supplement: drink ingestion; Behavioral: resistance-type exercise

INTERVENTIONS:
Dietary Supplement: drink ingestion — drink ingestion of a vanilla-flavoured beverage from a non-transparent shaker
  Other Names: supplement
Behavioral: resistance-type exercise — Lower body resistance-type exercise on the supine leg press and seated knee extension machine. Both machines 4 sets at 80% 1RM for 8-10 reps.
  Other Names: resistance training; strength training

SUMMARY:
Muscle tissue consists of proteins. These proteins are built up of small building blocks: amino acids. By consuming enough protein in our diet, we make sure that the body is provided with enough amino acids to facilitate muscle protein building. Also after exercise is protein intake important as it contributes to the recovery process. Providing the growing world population with sufficient animal-derived protein is a challenge. Plant proteins can be produced on a more sustainable commercial scale than conventional animal-derived proteins and therefore, can contribute to feeding our future population. Canola protein is a protein that is derived from rapeseed. The composition of canola seems to be comparable to that of other high-quality animal-based protein sources. But there is no data yet on the effect of canola protein ingestion on muscle growth. Additionally, most research on the effect of protein intake and muscle growth/recovery has been performed in males and we need more insight into the effect in females. The goal of this study is to investigate whether the ingestion of canola protein can stimulate muscle growth just as good as whey protein after a strength exercise session in females.

Primary objective: To assess the impact of 20g canola or 20g whey protein vs placebo ingestion on acute 5-hour postprandial muscle protein synthesis rates during recovery from lower-body resistance-type exercise in vivo in young females.

Secondary objective: To assess the impact of 20g canola protein vs 20g whey protein ingestion on acute 5-hour postprandial muscle protein synthesis rates during recovery from lower-body resistance-type exercise in vivo in young females.

Tertiary objectives: Compare signaling pathways and. postprandial 5-hour plasma glucose, insulin, and amino acid concentrations, (including area under the curve, peak concentrations, and time to peak) following canola protein, whey protein, and placebo ingestion during recovery from lower-body resistance-type exercise in young females.

Hypothesis: it is hypothesized that acute 5-hour postprandial muscle protein synthesis rates will be not different following 20g canola protein and 20g whey protein ingestion and higher compared to placebo during lower-body post-exercise recovery in healthy young females.

DETAILED DESCRIPTION:
Screening and pre-testing To assess whether volunteers are eligible to participate in this study, we will invite them to the University for a screening. At the start of the screening session, the entire experimental trial will be explained and any potential questions will be answered. Thereafter, the volunteers are asked to read, fill out, and sign the informed consent form. After signing the informed consent form, the participant's eligibility will be assessed based on the in- and exclusion criteria. To further assess their eligibility, participants will be asked to fill out a medical questionnaire to assess their general health, use of medication, habitual food intake, and physical activity (Appendix F1.1). Next, blood pressure will be assessed. Body mass (with accuracy of 0.1 kg) and height (with accuracy of 0.01 m) will be determined, and body composition will be assessed via a Dual Energy X-ray Absorptiometry (DEXA) scan. A DEXA scan is a simple, non-invasive procedure. At the beginning of the procedure, subjects will be asked to lie down on a scanning table wearing underwear and they need to remain motionless during the measurements. As the scanner moves, a dual energy beam passes through the targeted skeletal muscle section and is measured by a detector. This procedure is repeated until the whole body is scanned and takes approximately 3 minutes.

The screening sessions will take place in the morning and participants are instructed to not have any breakfast in the morning in order to avoid perturbations in the DEXA scan.

In the event of an unexpected medical finding during the screening, subjects will always be notified. If a subject does not want to receive this notification, she cannot participate in the study.

Next, subjects will be familiarized and tested for bilateral strength on the exercise machines. First, participants will warm up on a cycle ergometer for 5 minutes at 100W. Subjects will be instructed on proper weight-lifting technique on each exercise machine (leg-press and leg-extension) and complete a standardized testing protocol to determine a measurement of maximal strength (1RM) for each exercise machine. In short, subjects will be seated on a leg press and leg extension machine and start with a warm-up of 2 sets of 10 repetitions with self-chosen weights. Then the load will be increased above the warming-up weight. The load will be increased after each successful lift, until failure, to determine maximal strength. A repetition is classified as "valid" if the participant is able to complete the entire lift in a controlled manner, without assistance.

When the screening is successfully performed, the test day will be scheduled. In order to prevent major impact from the menstrual cycle on the measurements of protein metabolism, the test day will be scheduled to take place in the first 10 days of the follicular phase.

Each subject will participate in an experimental trial lasting ~9h. Subjects will be instructed to arrive at the university at 7:45 AM in an overnight fasted and rested state, meaning that participants are not allowed to eat and drink (except for water) from 22:00 the night prior to the experimental trial. They will be instructed to come to the university by car or public transportation. After the subjects arrive at the University, we will ask them to put on their shorts, determine their body mass, and assign them to a bed. Subjects will rest in a supine position and a Teflon catheter will be inserted in a heated dorsal hand vein and placed in a hot-box (60°C) for arterialized blood sampling. A baseline blood sample (Serum + plasma = 20 mL) will be collected at t= -210min to determine the amino acid enrichment level prior to the intervention. Following basal blood sample collection, a second Teflon catheter will be inserted into an antecubital vein of the contralateral arm for stable isotope infusion with the amino acids 13C6-phenylalanine and 2H2-tyrosine. At the start of the isotope infusion, the plasma phenylalanine and tyrosine pools will be primed with a single dose of the tracer solution, directly thereafter the continuous tracer infusion will commence.

During the entire experimental test day, the hand with the dorsal hand catheter will be pre-heated for 10 minutes prior to every blood draw in a hot box at 60°C to increase blood flow. This makes it easier to collect blood and minimizes nutrient exchange from blood into other tissues. Therefore, it allows us to collect nutrient-rich (arterialized) blood from a vein. Arterialized blood samples (10mL) will be collected at t = -180, -120, -60, and 0 min to assess plasma tracer enrichments during the tracer infusion in the resting overnight post-absorptive period. After a pre-infusion period of 30 minutes (t = -180), during which the tracer infusion reaches steady state, a first muscle biopsy will be taken from the m. vastus lateralis to determine the background enrichment. At t=-45 min, a resistance-type exercise session will be performed (40 minutes). Subsequently, at t= 0 min a second biopsy will be taken from the same leg in order to assess the basal muscle protein synthetic rate. Immediately after the second biopsy, subjects will ingest the assigned drink (20g canola or whey protein or a non-caloric placebo). Subjects will be instructed to consume the drink within ~5 min.

Upon drink ingestion, the stopwatch will be reset (t= 0 min), and arterialized blood samples (10 mL) will be collected at t = 30, 60, 90, 120, 180, 240, and 300 min during the post-prandial period to assess plasma amino acid profiles and enrichments. To determine postprandial muscle protein synthesis (MPS), another biopsy will be taken at t = 300 min following meal ingestion from the contra-lateral leg. The muscle biopsy at t = 300 min allows us to obtain physiological relevant information with regard to the duration of the anabolic response to protein intake over a commonly used 5h postprandial period. Collectively, with the obtained biopsies we can measure muscle protein synthesis in the resting state (-180 - 0 min) and entire postprandial period (0 - 300 min; main outcome).

During the test day, a total of 3 muscle biopsies will be taken through 3 separate incisions, 2 biopsies from the one leg and 1 biopsy from the other leg. In total 12 times blood samples will be taken during the test day, the first sample that will be collected will be 20mL the subsequent samples 10mL, for a total of 130mL. Additionally, gastro-intestinal (GI) symptoms will be assessed at t = -60, 30, and 180 minutes and palatability at t = 15 min by questionnaires

ELIGIBILITY:
Inclusion Criteria:

* Female sex
* Aged between 18 and 35 y inclusive
* BMI between 18.5 and 30 kg/m2

Exclusion Criteria:

* Intolerant to milk products
* Mustard allergy
* Participating in a structured (progressive) exercise program
* Smoking regularly
* Diagnosed GI tract disorders or diseases
* Diagnosed musculoskeletal disorders
* Diagnosed metabolic disorders (e.g. diabetes)
* Hypertension (blood pressure above 140/90 mmHg)
* Donated blood 3 months prior to test day
* Pregnant
* Using third generation oral contraceptives
* Use of any medications known to affect protein metabolism (i.e. corticosteroids, non-steroidal anti-inflammatories).
* Chronic use of gastric acid suppressing medication
* Chronic use of anti-coagulants
* Recent (<1 year) participation in amino acid tracer (L-[ring-13C6]-phenylalanine and L-[3,5-2H2]-tyrosine studies

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-03-20 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Postprandial muscle protein fractional synthesis rate | 0-5 hours
  Muscle protein synthesis rates are calculated using L-ring-13C6-phenylalanine tracer and provided as 1 integrated value over the specified timeframe using plasma as precursor.

SECONDARY OUTCOMES:
'basal' muscle protein fractional synthesis rate | -3 - 0 hours
  Muscle protein synthesis rates are calculated using L-ring-13C6-phenylalanine tracer and provided as 1 integrated value over the specified timeframe using plasma as precursor.
Plasma glucose concentrations | 0-5 hours
  Plasma glucose concentrations
Plasma insulin concentrations | 0-5 hours
  Plasma insulin concentrations
Plasma amino acids concentrations | 0-5 hours
  Plasma amino acids concentrations

OTHER OUTCOMES:
Age in years | baseline at screening
  Age in years reported by participants
bodymass in kg | baseline at screening
  scale
Height in m | baseline at screening
  stadiometer
BMI in kg/m^2 | baseline at screening
  calculated from height and body mass
Whole body lean mass in kg | baseline at screening
  dexa
Appendicular lean mass in kg | baseline at screening
  dexa
bodyfat% | baseline at screening
  dexa
Dietary macronutrient intake | 2 days prior to experimental trial day
  assessed by written dietary intake records
Maximal leg strength | baseline at screening
  1-Repetition-maximum assessed on leg press and knee extension
drink palatability | On experimental trial day directly after drink ingestion
  Assessed by a visual analogue scale after drink ingestion

CONTACTS AND LOCATIONS:
Overall Officials: Luc van Loon, PhD, Principal Investigator — Maastricht University
Locations (1):
- Maastricht University Medical Centre+, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Boot N, Hermans WJ, Kuin LM, Malowany JM, Hendriks FK, Warnke I, Senden JM, Overman A, Goessens JP, Zorenc A, Kornips E, Verdijk LB, van Loon LJ. Ingestion of 20 g Whey or Canola Protein Does Not Further Increase Muscle Protein Synthesis Rates During Recovery From Resistance Exercise In Healthy, Young Females. J Nutr. 2025 Dec;155(12):4123-4135. doi: 10.1016/j.tjnut.2025.10.018. Epub 2025 Oct 14. PMID 41101508